CLINICAL TRIAL: NCT03028597
Title: Using Values Affirmation to Reduce the Effects of Stereotype Threat on Hypertension Disparities: The Multicenter Randomized HYpertension and VALUEs (HYVALUE) Trial
Brief Title: The Multicenter Randomized HYpertension and VALUEs (HYVALUE) Trial
Acronym: HYVALUE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); University of Colorado, Boulder (Other); Kaiser Permanente (Other); Denver Health and Hospital Authority (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 16-0510; 1R01HL133343-01 (NIH)
Record Dates: First submitted 2017-01-17; First posted 2017-01-23 (Estimated); Last update posted 2023-01-27 (Actual); Status verified 2022-11

CONDITIONS: Hypertension
Keywords: Hypertension; Medication Adherence; Values Affirmation; African Americans
MeSH Terms: conditions — Hypertension; Medication Adherence

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Values Affirmation (Experimental): The task first asks patients to reflect on a list of 11 personal values or self-defining skills.
  Interventions: Behavioral: Intervention Values Affirmation
- Control Values Affirmation (Active Comparator): The task first asks patients to reflect on a list of 11 personal values or self-defining skills.
  Interventions: Behavioral: Control Values Affirmation

INTERVENTIONS:
Behavioral: Intervention Values Affirmation — Participants are asked to circle the two or three values that are MOST important to them. Next, participants are asked to think about times when the values chosen might be important to THEMSELVES and then write a few sentences to describe when and why they might be important.
  Arms: Intervention Values Affirmation
Behavioral: Control Values Affirmation — Participants are asked to circle the two or three items that are LEAST important to them. Next, participants are asked to think about times when the values chosen might be important to SOMEONE ELSE and then write a few sentences to describe when and why they might be important.
  Arms: Control Values Affirmation

SUMMARY:
The objective of this study is to reduce the effects of stereotype threat on the adherence of African American patients with hypertension.

The specific aims of this study, which employs a values affirmation intervention, are to:

1. Compare the effects of the values-affirmation exercise to a control condition on antihypertensive medication adherence in African American patients with uncontrolled hypertension across three clinical settings,
2. Compare the effects of the values-affirmation exercise on antihypertensive medication adherence in African American patients and white patients with uncontrolled hypertension and similar socioeconomic characteristics, and
3. Evaluate the intervention for widespread dissemination using the RE-AIM (reach, effectiveness, adoption, implementation and maintenance) framework

DETAILED DESCRIPTION:
One in 3 US adults has hypertension and African Americans are disproportionately affected; almost 40% of non-Hispanic blacks have hypertension. Although the rates of uncontrolled hypertension have been decreasing in all groups, African Americans continue to have higher rates of uncontrolled hypertension compared to white Americans. The Institute of Medicine, World Health Organization and others have identified poor adherence to medications as the most significant, modifiable contributor to uncontrolled hypertension.

Stereotype threat may contribute to low adherence. Stereotype threat occurs when cues in the environment (such as visiting a doctor's office) trigger the threat of confirming, as self-characteristic, a negative stereotype about one's group. Although any individual may experience stereotype threat, African Americans are at greater risk due to widespread racism and past experiences of discrimination.

Values affirmation interventions reduce stereotype threat and decrease racial disparities in various outcomes. Values affirmation exercises typically ask participants to write a few sentences about their core values. By focusing on values that are important to them, values affirmation bolsters a person's self-concept by helping them view themselves as adequate, effective, and able to control important outcomes in spite of a possible threat.

Based on the evidence supporting the effectiveness of values affirmation in educational and other settings, the investigators hypothesize that values affirmation can similarly reduce racial disparities in medication adherence and subsequent health outcomes. By asking participating intervention patients to engage in a values affirmation exercise at an initial appointment with a primary care provider, the investigators hope to improve hypertensive medication adherence, systolic blood pressure, time under blood pressure control, and treatment intensification, and to reduce racial disparities in these outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Hypertension diagnosis: primary or secondary ICD-10 code diagnosis in last 24 mo
* SBP >140 mm Hg or DBP >90 mm Hg in last 12 months
* Currently taking antihypertensive medications
* Medications filled within health system's pharmacy
* White or African American, self-reported race
* Upcoming primary care visit
* Ability to read and write English

Exclusion Criteria:

* Pregnancy-related hypertension
* Dialysis-dependent end-stage renal disease
* Prisoners
* Unable to provide consent

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 960 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2021-05 (Actual); Study Completion 2021-05 (Actual)

PRIMARY OUTCOMES:
Change in Antihypertensive Medication Adherence using Pharmacy Records | Baseline, 3 and 6 months
  This antihypertensive medication adherence outcome will be a summary measure of adherence which assesses the proportion of days covered (PDC) over the period of observation for which a patient obtains antihypertensive medications. Adherence will be calculated for each antihypertensive drug in the regimen and combined across drugs into a summary measure of adherence for the entire drug regimen.
Change in Antihypertensive Medication Adherence using Self-Reported Adherence | Baseline, 3 and 6 months
  This antihypertensive medication adherence outcome will be a summary measure of self-reported adherence using the validated Voils instrument, which has 3 questions that address adherence over the previous 7 days.
Change in Antihypertensive Medication Adherence using Pill Counts | Baseline, 3 and 6 months
  This antihypertensive medication adherence outcome will be a summary outcome measure of adherence where if x is the number of pills in the bottle, y is the number of pills that would have been in the bottle had all pills been taken since the bottle was filled, and z is the number of pills that should have been taken since the last fill, and adherence is calculated as 1- [(x-y)/z].

SECONDARY OUTCOMES:
Systolic Blood Pressure | Baseline, 3 and 6 months
  Systolic blood pressure over time
Proportion of Time Blood Pressure is Under Control | 6 months
  Defined as the proportion of time over the 6-months of follow-up with a BP ≤ 140/90 mmHg.
Average Treatment Intensification | 6 months
  Calculated by subtracting the number of expected intensifications (number of visits after enrollment with a BP ≥140/90 mm Hg) from the number of observed intensifications (either an increase in dose or addition of a new medication class), and then dividing this difference by the number of office visits over the observation period.

CONTACTS AND LOCATIONS:
Overall Officials: Stacie L Daugherty, MD, MSPH, Principal Investigator — University of Colorado, Denver
Locations (3):
- United States (3):
  - Denver Health and Hospital Authority, Denver, Colorado
  - Kaiser Permanente of Colorado, Denver, Colorado
  - Kaiser Permanente Mid Atlantic States, Rockville, Maryland

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD at this time.

REFERENCES:
- [Derived] Gust CJ, Bryan AD, Havranek EP, Vupputuri S, Steiner JF, Blair IV, Hanratty R, Daugherty SL. Health Behavior Theory and Hypertension Management: Comparisons Among Black, White, and American Indian and Alaska Native Patients. Race Soc Probl. 2022 Dec;14(4):369-382. doi: 10.1007/s12552-022-09359-2. Epub 2022 Feb 25. PMID 38322707
- [Derived] Genelin MP, Helmkamp LJ, Steiner JF, Maertens JA, Hanratty R, Vupputuri S, Havranek EP, Dickinson LM, Blair IV, Daugherty SL. Patient Pill Organization Strategies and Adherence Measured in a Cross-Sectional Study of Hypertension. Patient Prefer Adherence. 2023 Mar 23;17:817-826. doi: 10.2147/PPA.S399693. eCollection 2023. PMID 36992865
- [Derived] Henderson KH, Helmkamp LJ, Steiner JF, Havranek EP, Vupputuri SX, Hanratty R, Blair IV, Maertens JA, Dickinson M, Daugherty SL. Relationship Between Social Vulnerability Indicators and Trial Participant Attrition: Findings From the HYVALUE Trial. Circ Cardiovasc Qual Outcomes. 2022 May;15(5):e007709. doi: 10.1161/CIRCOUTCOMES.120.007709. Epub 2022 Apr 14. PMID 35418247
- [Derived] Daugherty SL, Helmkamp L, Vupputuri S, Hanratty R, Steiner JF, Blair IV, Dickinson LM, Maertens JA, Havranek EP. Effect of Values Affirmation on Reducing Racial Differences in Adherence to Hypertension Medication: The HYVALUE Randomized Clinical Trial. JAMA Netw Open. 2021 Dec 1;4(12):e2139533. doi: 10.1001/jamanetworkopen.2021.39533. PMID 34913976
- [Derived] Daugherty SL, Vupputuri S, Hanratty R, Steiner JF, Maertens JA, Blair IV, Dickinson LM, Helmkamp L, Havranek EP. Using Values Affirmation to Reduce the Effects of Stereotype Threat on Hypertension Disparities: Protocol for the Multicenter Randomized Hypertension and Values (HYVALUE) Trial. JMIR Res Protoc. 2019 Mar 25;8(3):e12498. doi: 10.2196/12498. PMID 30907744